CLINICAL TRIAL: NCT05408715
Title: An International Prospective Natural History Study in Children With a Type II Collagen Disorder With Short Stature
Brief Title: A Natural History Study in Children With a Type II Collagen Disorder With Short Stature
Acronym: ROCKET
Status: Recruiting | Type: Observational
Sponsor: Innoskel (Industry)
Responsible Party: Sponsor
Other Study IDs: COL221-101
Record Dates: First submitted 2022-05-13; First posted 2022-06-07 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: SEDC; Hypochondrogenesis; Semd, Strudwick Type; Kniest Dysplasia
Keywords: Skeletal Dysplasia; Short Stature; Bone Disease
MeSH Terms: conditions — Hypochondrogenesis; Strudwick syndrome; Kniest dysplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood (5-10 ml) will be collected to measure biomarkers related to bone growth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Natural History Study — Longitudinal assessment of symptoms and development of complications in type II collagen disorders

SUMMARY:
There are relatively few data available on type II collagen disorders, and evidence is lacking on the disease course in relation to symptoms and development of complications, the level of actual disease burden over time as well as data to support identification of possible risk factors.

This study aims to build a natural history data set through collection of a number of clinical, imaging, and laboratory assessments that may be specific predictors of type II collagen disorder progression and clinical outcome. Having a type II collagen disorder natural history data set can inform potential efficacy endpoints and biomarkers for future clinical trials.

This natural history study will follow up to 60 individuals diagnosed with a type II collagen disorder for up to 3 years. Visits will be conducted every 3 months for the first year and then every 6 months, during which several assessments will be performed in order to learn about the natural course of the disease, including changes in clinical and functional outcomes, imaging and biofluid biomarkers. Some of the study activities include: a physical exam, height measurements, vision and breathing tests and x-ray. A blood sample will be collected once or twice each year.

Most of the information collected, the tests done, and the schedule of visits in this study are the same as recommended for regular care of children with a type II collagen disorder.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type II collagen disorder with short stature at birth (2 standard deviations (SD) or more below the mean) i.e., Hypochondrogenesis, Kniest, Spondyloepiphyseal dysplasia congenita (SEDc) Spondyloepimetaphyseal dysplasia (SEMD) Strudwick type, Spondyloperipheral dysplasia (SED).
* Children up to and including 12 years of age, up to the day before their 13th birthday, on the date of consent/assent.
* The patient is sufficiently able, in the opinion of the Investigator, to adhere to the study visit schedule and other protocol requirements.
* The patient's parent(s) or legal guardian(s) has signed written informed consent, according to the local regulations and after all relevant aspects of the study have been explained and discussed.
* The child (depending on local institutional review board/ethical committee requirements) has provided assent.

Exclusion Criteria:

* Tanner stage 3 or more based on investigator assessment during physical examination
* The patient has a diagnosis of any short stature condition other than a type II collagen disorder.
* The investigator and/or clinical study advisory committee considers the patient has a type II collagen disorder which is not Hypochondrogenesis, SEDc, Kniest, SEMD or SED i.e., Stickler.
* The patient has any other medical condition that may impact growth or where the treatment is known to impact growth, such as but not limited to hypothyroidism or hyperthyroidism, insulin-requiring diabetes mellitus, autoimmune inflammatory disease, autonomic neuropathy or inflammatory bowel disease.
* Treatment in the previous 12 months prior to consent/assent with growth hormones, insulin-like growth factor 1, anabolic steroids, or any other drug expected to affect growth velocity. Brief (up to a few weeks) use of steroids is permitted.
* Participation in any interventional clinical trial or treatment for a type II collagenopathy.
* Has any condition or circumstance that in the view of the investigator places the child at high risk of poor compliance with the visit schedule or of not completing the study.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and children with a type II collagen disorder with short stature from birth to 12 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of relevant medical data (retrospective and prospective) | Up to 3 years
  Collection of demographic data, collagen type II-related medical complications, past medical and surgical history and current medication.
Anthropometric measurements | Up to 3 years
  Collection of consistent growth measurements (in centimeters).
Change over time in motor function in children 2 years old and younger | Up to 2 years
  Motor development will be assessed using the World Health Organisation (WHO) Motor Milestones.
Change over time in motor function in children >2 years old | Up to 3 years
  Timed 100-meter walk/run test (T100T). In the T100T, the participant is instructed to walk as fast as possible for a distance of 100 meters. Timed 10-meter walk/run test (T10T). Participants walk 10-meters at self-selected pace. Functional Mobility Scale (FMS) rates the walking ability in three different walking distances.
Change over time in pulmonary function | Up to 3 years
  Lung function measured through spirometry in all participants >4 years of age
Change over time in ophthalmological assessment | Up to 3 years
  Standard ophthalmological assessment.
Change over time in skeletal abnormalities | Up to 3 years
  Investigators should collect radiographs according standard of care to determine change in skeletal abnormalities and bone growth.
Measurement of biomarkers for bone growth | Up to 3 years
  Changes from baseline in serum collagen X fragments.
Measurement of CNP/ProCNP | Up to 3 years
  Changes from baseline in serum CNP/ProCNP
Measurement of bone-specific alkaline phosphatase (BALP) | Up to 3 years
  Changes from baseline in serum BALP
Change in scores for the pediatric quality of life inventory parent report (PedsQL) | Up to 3 years
  The PedsQL parent-proxy report has 23 items that investigate physical, emotional, and social QoL as well as school functioning.
Change in PROMIS pediatric short form pain behaviors score | Up to 3 years
  The PROMIS pediatric short form pain behaviors, parent-proxy report is an 8-item measure completed by parents that assesses pain behaviors displayed by their child in the past 7 days. Total scores are standardized to a T-score with a mean of 50 and a standard deviation of 10, where higher scores indicate increased behaviors due to pain.
Change in fatigue | Up to 3 years
  The PROMIS pediatric fatigue parent-proxy report is completed by parents to assess their child's ability to carry out daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Superti-Furga, Principal Investigator — Centre hospitalier universitaire vaudois, Lausanne
Locations (2):
- Hopital Necker-Enfants Malades, Paris, France
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Savarirayan R, Bompadre V, Bober MB, Cho TJ, Goldberg MJ, Hoover-Fong J, Irving M, Kamps SE, Mackenzie WG, Raggio C, Spencer SS, White KK; Skeletal Dysplasia Management Consortium. Best practice guidelines regarding diagnosis and management of patients with type II collagen disorders. Genet Med. 2019 Sep;21(9):2070-2080. doi: 10.1038/s41436-019-0446-9. Epub 2019 Jan 30. PMID 30696995
- [Background] Oh CW, Thacker MM, Mackenzie WG, Riddle EC. Coxa vara: a novel measurement technique in skeletal dysplasias. Clin Orthop Relat Res. 2006 Jun;447:125-31. doi: 10.1097/01.blo.0000203476.81302.24. PMID 16505708
- [Background] Dhiman N, Albaghdadi A, Zogg CK, Sharma M, Hoover-Fong JE, Ain MC, Haider AH. Factors associated with health-related quality of life (HRQOL) in adults with short stature skeletal dysplasias. Qual Life Res. 2017 May;26(5):1337-1348. doi: 10.1007/s11136-016-1455-7. Epub 2016 Nov 19. PMID 27866314
- [Background] Graham HK, Harvey A, Rodda J, Nattrass GR, Pirpiris M. The Functional Mobility Scale (FMS). J Pediatr Orthop. 2004 Sep-Oct;24(5):514-20. doi: 10.1097/00004694-200409000-00011. PMID 15308901